CLINICAL TRIAL: NCT00675363
Title: A Randomized Trial of Daily Sedative Interruption in Critically Ill, Mechanically Ventilated Patients Being Managed With a Sedation Protocol
Brief Title: Daily Sedative Interruption in Critically Ill Patients Being Managed With a Sedation Protocol.
Acronym: SLEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Sangeeta Mehta, M.D., Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 85487
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2018-03

CONDITIONS: Critical Illness
Keywords: ICU; Sedation strategies; Daily sedative interruption; Sedation protocols; Mechanical Ventilation; Sedation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PS (Active Comparator): Nurse-directed protocols for administering sedation and/or analgesia by continuous infusion.
  Interventions: Procedure: Protocolized Sedation
- PS + DI (Active Comparator): Nurse-directed protocols for administering sedation and/or analgesia, with daily interruption of sedation/analgesia
  Interventions: Procedure: Protocolized sedation, with daily interruption

INTERVENTIONS:
Procedure: Protocolized Sedation — Nurse-directed protocol for administering sedation and/or analgesia.
  Arms: PS
Procedure: Protocolized sedation, with daily interruption — Nurse-directed protocols for administering sedation and/or analgesia, with daily interruption of sedation/analgesia
  Arms: PS + DI

SUMMARY:
The purpose of this study is to determine whether the use of both a nurse-driven sedation protocol and daily sedative interruption, compared with a sedation protocol alone, result in better outcomes for mechanically ventilated adults.

DETAILED DESCRIPTION:
All critically ill, mechanically ventilated patients in the Intensive Care Unit receive medications to relieve pain and anxiety. However, accumulation of these medications can be associated with serious complications, most notably longer time on the breathing machine and in the ICU. Two strategies have been shown to dramatically improve patient outcomes: nurse-directed protocols for giving sedation, and daily interruption of sedation. However, these strategies have not been widely adopted, because of physicians' concerns, and because it is unclear which strategy is better. Given that patient outcome is improved with either of these strategies, the fundamental question that arises is whether patients managed with a combination of two strategies which both reduce drug accumulation (protocolized sedation and daily interruption) have an even better outcome than patients managed with only one of them (protocolized sedation).We are conducting a multicenter randomized trial in which 400 critically ill, mechanically ventilated patients will have their sedation managed with protocolized sedation alone, or both strategies. Primary outcomes are duration of mechanical ventilation and ICU and hospital lengths of stay. Secondary outcomes are the incidence of delirium, the use of neurologic tests, nurse and respiratory therapist effort associated with the sedation management, the incidence of patient self-removal of lines and tubes, and patient recall of the ICU stay. The results of this large multi-center trial will help to inform best practice with regard to sedation management of critically ill patients in Canada and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Mechanically ventilated, with anticipated need for MV ≥48 hrs
* ICU team has decided to initiate continuous sedative/analgesic infusion(s)
* informed consent from patient and/or SDM

Exclusion Criteria

* Admission after resuscitation from cardiac arrest
* Traumatic brain injury
* Currently receiving neuromuscular blocking agents
* Allergy to midazolam and lorazepam
* Lack of commitment to aggressive treatment
* Previous enrolment in SLEAP, or current enrolment in related trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2012-10-17 (Actual)

PRIMARY OUTCOMES:
time to successful extubation | This will be the length of time that the patient remains on continuous infusions of sedation and/or analgesia in the ICU. At 60 days, all study interventions will terminate, but patients will be followed for outcomes.

SECONDARY OUTCOMES:
ICU and hospital lengths of stay, ICU and hospital mortality, Adverse events (e.g., self -removal of endotracheal tube) | This will be the length of time that the patient remains on continuous infusions of sedation and/or analgesia in the ICU. At 60 days, all study interventions will terminate, but patients will be followed for outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Mehta, M.D., Principal Investigator — MOUNT SINAI HOSPITAL
Locations (16):
- United States (2):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Tuft's Medical Centre, Boston, Massachusetts
- Canada (14):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Vancouver, British Columbia
  - Providence Health Care-St. Paul's Hospital, Vancouver, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joesph's Healthcare, Hamilton, Ontario
  - Sunnybrook HSC, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Maisonneuve Rosemount, Montreal, Quebec

REFERENCES:
- [Derived] Mehta S, Meade M, Burry L, Mallick R, Katsios C, Fergusson D, Dodek P, Burns K, Herridge M, Devlin JW, Tanios M, Fowler R, Jacka M, Skrobik Y, Olafson K, Cook D; SLEAP Investigators and the Canadian Critical Care Trials Group. Variation in diurnal sedation in mechanically ventilated patients who are managed with a sedation protocol alone or a sedation protocol and daily interruption. Crit Care. 2016 Aug 1;20(1):233. doi: 10.1186/s13054-016-1405-3. PMID 27480314
- [Derived] Rose L, Burry L, Mallick R, Luk E, Cook D, Fergusson D, Dodek P, Burns K, Granton J, Ferguson N, Devlin JW, Steinberg M, Keenan S, Reynolds S, Tanios M, Fowler RA, Jacka M, Olafson K, Skrobik Y, Mehta S. Prevalence, risk factors, and outcomes associated with physical restraint use in mechanically ventilated adults. J Crit Care. 2016 Feb;31(1):31-5. doi: 10.1016/j.jcrc.2015.09.011. Epub 2015 Sep 25. PMID 26489482
- [Derived] Burry L, Cook D, Herridge M, Devlin JW, Fergusson D, Meade M, Steinberg M, Skrobik Y, Olafson K, Burns K, Dodek P, Granton J, Ferguson N, Jacka M, Tanios M, Fowler R, Reynolds S, Keenan S, Mallick R, Mehta S; SLEAP Investigators; Canadian Critical Care Trials Group. Recall of ICU Stay in Patients Managed With a Sedation Protocol or a Sedation Protocol With Daily Interruption. Crit Care Med. 2015 Oct;43(10):2180-90. doi: 10.1097/CCM.0000000000001196. PMID 26181221
- [Derived] Rose L, Fitzgerald E, Cook D, Kim S, Steinberg M, Devlin JW, Ashley BJ, Dodek P, Smith O, Poretta K, Lee Y, Burns K, Harvey J, Skrobik Y, Fergusson D, Meade M, Kraguljac A, Burry L, Mehta S; SLEAP Investigators; Canadian Critical Care Trials Group. Clinician perspectives on protocols designed to minimize sedation. J Crit Care. 2015 Apr;30(2):348-52. doi: 10.1016/j.jcrc.2014.10.021. Epub 2014 Oct 30. PMID 25466317
- [Derived] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503